CLINICAL TRIAL: NCT07380503
Title: Analgesic Efficacy of Adding Different Doses of Dexmedetomidine as Adjuvants With Bupivacaine vs.Bupivacaine Only in Ultrasound-guided Erector Spinae Plane Block in Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery. A Randomized Controlled Double Blinded Study.
Brief Title: Different Doses of Dexmedetomidine With Bupivacaine vs.Bupivacaine Only in Ultrasound-guided Erector Spinae Plane Block in Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Ahmed Abdalla Mohamed Ali Nasr (Unknown); Dina Soliman Mohammed Idris (Unknown); Mohamed Nabil Elshafie Abdulkader (Unknown); Mohamed Ahmed Abd El Hamed Shamma (Unknown); Aya Sayed Ali Ahmed Mostafa (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia&Surgical ICU and Pain Clinic, Cairo University
Other Study IDs: MD-402-2024
Record Dates: First submitted 2025-11-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: ESPB With Dexmetomidine May Provide Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 (ESPB alone): The block was performed with full aseptic precautions. A convex ultrasound probe was wrapped in a sterile lens sleeve, and the sagittal side position of the probe (approximately 3 cm) was used to locate the bilateral T7 transverse process. We used an in-plane needle technique, inserting a 21-gauge needle (Sonoplex cannula)+ into the surface of the transverse process in a caudal to cranial direction. There was no blood or cerebrospinal fluid while withdrawing the syringe plunger. Saline (3 mL) was injected between the erector spinae muscle and the transverse process for hydrodissection to confirm the correct position., 20 mL of 0.25% bupivacaine was administered between the erector spine muscle and transverse process.
  Local anesthetic diffusion between the transverse process and erector spine muscle is an indication of a successful puncture.
  Interventions: Drug: Analgesic Efficacy of adding different doses of dexmedetomidine
- Group 2 (ESPB with dexamedatomedine 1 mcg/kg): The erectospinae plane block was performed bilaterally with 20 ml 0.25 % bupivacaine prepared as follows: 10 ml bupivacaine 0.5% + 1 mcg per kg dexmedatomidine (2ml)+ 8 ml normal saline
  Interventions: Drug: Analgesic Efficacy of adding different doses of dexmedetomidine
- Group 3 (ESPB with dexamedatomedine (1.5 mcg/kg): The erectospinae plane block was performed bilaterally with 20 ml 0.25 % bupivacaine prepared as follows: 10 ml bupivacaine 0.5% + 1.5 mcg per kg dexmedatomidine (2ml)+ 8 ml normal saline
  Interventions: Drug: Analgesic Efficacy of adding different doses of dexmedetomidine

INTERVENTIONS:
Drug: Analgesic Efficacy of adding different doses of dexmedetomidine — Analgesic Efficacy of adding different doses of dexmedetomidine as adjuvants with bupivacaine vs. bupivacaine

SUMMARY:
Analgesic Efficacy of adding different doses of dexmedetomidine as adjuvants with bupivacaine vs. bupivacaine only in ultrasound-guided erector spinae plane block in morbidly obese patients undergoing Laparoscopic Bariatric surgery. A RANDOMIZED CONTROLLED DOUBLE BLINDED STUDY.

DETAILED DESCRIPTION:
Bariatric surgery is recognized as an essential and effective treatment for obesity and relevant metabolic diseases, such as type 2 diabetes . With the promotion of enhanced recovery after surgery (ERAS) in bariatric surgery, the administration of the ERAS protocol has been widely accepted . Compared with traditional treatment, ERAS reduces the potential opportunity for postoperative complications, ultimately improving the quality of care for patients . Inadequate postoperative pain management for patients may increase the amount of opioid analgesic drugs consumed, prolong time to off-bed activity and hospitalization, augment the incidence of relevant complications, increase medical costs, and reduce the quality of life Laparoscopic bariatric surgeries are considered minimally invasive procedures, but they can cause severe pain . Opioids are excellent analgesics, but they have many side effects as respiratory depression, which may further complicate pain management in bariatric surgeries, particularly in cases with obstructive sleep apnea . Other comorbidities such as diabetes mellitus and cardiovascular diseases that are common in patients with obesity can also lead to difficulties with pain management . This complexity highlights the challenges of the optimal choice of analgesia in bariatric surgery.

The new regional blocking technique (Erector spinae plane block) can utilize to reduce postoperative pain effectively in various surgical procedures such as breast, thoracic, abdominal and lumbar surgery . However, although usually the use of long-acting local anesthetics (LAs), not provide long duration of action . Even though continuous catheter-based nerve block can prolong the postoperative pain relief time, this technique requires additional time and cost, and increases the risk of infection and neurological complications Dexmedetomidine (DEX) is a highly selective alpha-2 adrenergic receptor agonist with sedative and analgesic sparing effects, reduced delirium and agitation, with additive perioperative sympatholysis, cardiovascular stabilizing effects, and preservation of respiratory function..

In previous clinical studies, DEX as adjuvant to LAs as the potential to prolong blockade duration. However, it remains unclear whether Dex as an adjunct for bupivicaine to ESPB can significantly improve the quality of postoperative analgesia and recovery after Laproscopic bariatric surgery in morbidly obese patients. Thus, the main objective of the present study was to explore the effects of different dosages of Dex as an adjunct for bupivicaine combined with ESPB on the quality of postoperative analgesia and recovery and achieve opioid free anasthesia in patients following laproscopic bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* Age starting from 21 to 60 years.
* Genders eligible for study: Male and female sexes.
* ASA I-III
* Undergoing Laparoscopic bariatric surgery.
* BMI > = 40.

Exclusion Criteria:

* Patient refusal
* Known allergy to local anesthetics and adjuvant drugs used (dexamedatomedine)
* Bleeding disorders; platelets count <50,000, prothrombin concentration < 60% or any coagulopathy disorder.
* Use of any anti-coagulants
* Inability to provide informed consent
* ASA -IV
* Neurological disorders
* Patient with psychiatric disorders
* Failed block is claimed if the patient required more than 2 doses of rescue analgesia in the first 2 hrs post operative , failed block cases will be recorded , excluded and managed according to the institutional regulations (opioid analgesia).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Patients were assessed the day before surgery in a preoperative visit for evaluation of their medical status, laboratory investigations and for fulfilling all the above inclusion and exclusion criteria. 20g cannula inserted in holding area. Premedication with 0.02 mg/kg midazolam was administered intravenously 5 minutes before block performance.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption in Day 1 | Day 1
  Postoperative opioid consumption in Day 1

SECONDARY OUTCOMES:
Visual Analogue Scale | Ffirst day
  Visual Analogue Scale (VAS) pain score assessed immediately postoperatively and then at 30 minutes, 1, 2, 4, 6, 12 and 24 h. Scores (1-3) were considered mild pain, (4-6) moderate pain and (7-10) severe pain
Time to first postoperative rescue analgesia | Time to first postoperative rescue analgesia in one day
  Total dose of fentanyl required intraoperative (including induction dose) to be 200 microgram
Ramzy sedation score: | Day 1
  * Score 1:Awake;agitated or restless or both.
  * Score 2: Awake; cooperative, oriented and tranquil.
  * Score 3: Awake but responds to commands only
  * Sore 4: Asleep; brisk response to light glabellar tap or loud auditory stimulus.
  * Score 5: Asleep; sluggish response to light glabellar tap or loud auditory stimulus
  * Score 6: Asleep; no response to glabellar tap or loud auditory stimulus
Effect on arterial blood pressure | Day 1
  Effect on arterial blood pressure
Number and percentage of people developing side effects of block (pneumothorax, vascular injury). | Day 1
  Number and percentage of people developing side effects of block (pneumothorax, vascular injury).
Number and percentage of side effects related to adjuvant drugs as bradycardia and hypotension. | Through Study Completion
  Number and percentage of side effects related to adjuvant drugs as bradycardia and hypotension.
Local anesthetic toxicity. | Through Study Completion
  Local anesthetic toxicity
Post operative nausea and vomiting. | Through Study Completion
  Post operative nausea and vomiting.
Effect on heart rate | Day 1
  Effect on heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
When study completed